CLINICAL TRIAL: NCT01057420
Title: Effect of Hyperoxemia on Platelet Function in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Johannes Wacker, MD, Surgical Intensive Care Medicine, UniversitaetsSpital Zurich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: O2Tc-2009
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhalation of 80% Oxygen (Other): Inhalation of 80% Oxygen by nonrebreathing reservoir face masks for 4 hours
  Interventions: Drug: oxygen inhalation

INTERVENTIONS:
Drug: oxygen inhalation — Inhalation of 80% oxygen via face mask

SUMMARY:
Prospective, controlled, randomized crossover volunteer study to investigate the effect of hyperoxemia due to inhalation of oxygen (80% inspiratory fraction) via reservoir-face-mask on blood coagulation, especially platelet function, as measured by thrombelastography. According to results of basic animal and in vitro investigations, hyperoxemia may activate platelets by means of reactive oxygen species. This study aims at investigating a possible pro-coagulant effect of hyperoxemia in healthy volunteers. Additional studies on possible mechanisms are integrated.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* informed consent; no coagulation disorder or other illnesses;
* non-smoker;
* women: no pharmacological contraception, negative pregnancy test;
* 25-45 years old; no medication; no acute or chronic airway problems;
* for 24 hours before study: no extreme physical activity, no polyphenol-containing food (red wine, apples, cabbage, garlic);
* for 48 hours: no caffeine-containing drinks, no dark chocolate.

Exclusion criteria:

* Lack of one of the inclusion criteria;
* allergy or incompatibility to substances/materials applied in the study;
* very thin veins/arteries.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
maximum amplitude in thrombelastography | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Wacker, MD, Principal Investigator — Surgical Intensive Care Medicine, UniversitaetsSpital Zuerich; Reto Stocker, Prof., MD, Study Director — Surgical Intensive Care Medicine, UniversitaetsSpital Zurich
Locations (1):
- Surgical Intensive Care Medicine, Zurich, Switzerland